CLINICAL TRIAL: NCT04690920
Title: Theranostic Implication of Complimentary Medicines Against IL-6/Gp-130 in COVID-19.: An in Vitro and in Silco Approach
Brief Title: Theranostic Implication of Complementary Medicines Against Interleukin Receptors and Gp-130 Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Dr Muhammad Mansoor Hafeez, Doctor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOL/IMBB/2020/118
Record Dates: First submitted 2020-12-19; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Corona Virus Disease 2019 (COVID-19)
Keywords: corona virus disease 2019 (COVID-19); Tocilizumab; Remdesivir; Interleukin receptor-6, glycoprotein-130; receptor blocker
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab; remdesivir; Anti-Bacterial Agents; Oxygen; Ascorbic Acid; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention)
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab
- Remdesivir (Experimental)
  Interventions: Drug: Tocilizumab
- Standard Treatment (Active Comparator)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Comparison of drugs, Tocilizumab, Remdesivir, standard treatment with controls
  Other Names: Remdesivir; Standard treatment with Antibiotic, oxygen, Vitamin C, Statins; No treatment is given to control group
  Arms: Remdesivir; Standard Treatment; Tocilizumab

SUMMARY:
IL-6 is an inflammatory marker, secrete by the cells in many pathological conditions like COVID-19 pneumonia. Interleukin 6 bind with its receptors (IL-6R) on cells surface and recruited a protein for its activation known as gp-130. Activated receptors send signals to nucleus through secondary messenger system and up regulate the expression of IL-6/GP130 domain. Total of two hundred (n=200) participants were included in the current study and divided equally in four groups. Group B is given Tocilizumab and Group C is treated with Remdesivir along with the approved standard treatment. Group D is only Given standard therapy and Group A constituted normal healthy age and sexed matched participants. Levels of gp-130 were estimated by commercially available ELISA kit. To estimate the relationship of severity of disease with gp-130 and IL-6 Pearson's correlations was used. Sensitivity and specificity for what purpose

ELIGIBILITY:
Inclusion Criteria:

Admitted diagnosed cases of COVID-19 infection on real time polymerase chain reaction (RT-PCR) Both male and female were included All participants were on oxygen therapy

Exclusion Criteria:

Asthmatics pulmonary fibrosis chronic obstructive pulmonary disease (COPD) Allergic to remdesivir Allergic to Actemra Refused to take consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male and female diagnosed as COVID-19 infected by polymerase chain reaction (PCR)
Enrollment: 200 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Ratio of partial pressure of oxygen in arterial blood to fraction of inhaled oxygen | 7 days

SECONDARY OUTCOMES:
Hospital stay | 15 days
Oxygen demand | 7-15 days
Viral load | 7-15 days
  by RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Arif Malik, PhD, Study Director — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
statistical analysis, results